CLINICAL TRIAL: NCT06480422
Title: Combined Effects Of Autogenic Drainage and Segmental Breathing Techniques in Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0381
Record Dates: First submitted 2024-06-11; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Autogenic Drainage,; Segmental breathing technique; Chronic Obstructive Pulmonary Disease.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- segmental breathing technique + Autogenic drainage (Experimental): For Segmental Breathing instruction, the therapist's hand is placed on the chest area to be expanded. The patient is encouraged to deeply breath and to preferentially "Send Air"to that area of chest where tactile stimulation is being applied by the therapist. On full expiration moderate compression is applied. To begin an autogenic drainage sit in a relaxed seated position with neck extended slightly. Blow patient's nose and huff, cough to clear your upper airways to mucus. This technique has three phases. Moving mucus from small airways (Unsticking), Moving mucus from small airways to medium sized airways(Collecting), Moving mucus from medium sized airways to large airways (Evacuation) Take in a deep breath. Hold the breath for three seconds. With some gentle force exhale all the air out of your lungs. Repeat three times. Do not cough untill after the third breath. Repeat sessions 3 times in a week for 4 almost weeks.
  Interventions: Other: Segmental breathing technique; Other: autogenic drainage
- Autogenic drainage (Active Comparator): To begin an autogenic drainage sit in a relaxed seated position with neck extended slightly. Blow ptient's nose and huff, cough to clear your upper airways to mucus.This technique has three phases. Moving mucus from small airways (Unsticking), Moving mucus from small airways to medium sized airways(Collecting), Moving mucus from medium sized airways to large airways(Evacuation) Take in a deep breath.Hold the breath for three seconds.With some gentle force exhale all the air out of your lungs. Repeat three times.Do not cough untill after the third breath.
  Repeat sessions 3 times in a week for 4 almost weeks.
  Interventions: Other: autogenic drainage

INTERVENTIONS:
Other: Segmental breathing technique — To begin an autogenic drainage sit in a relaxed seated position with neck extended slightly. Blow patient's nose and huff, cough to clear your upper airways to mucus. This technique has three phases. Moving mucus from small airways (Unsticking), Moving mucus from small airways to medium sized airways(Collecting), Moving mucus from medium sized airways to large airways(Evacuation) Take in a deep breath. Hold the breath for three seconds. With some gentle force exhale all the air out of your lungs. Repeat three times. Do not cough untill after the third breath. Repeat sessions 3 times in a week for 4 almost weeks. Repeat the cycle untill you have cleared your lungs as much as possible, 20 and 45 minutes.
  Other Names: Autogenic drainage
  Arms: segmental breathing technique + Autogenic drainage
Other: autogenic drainage — To begin an autogenic drainage sit in a relaxed seated position with neck extended slightly.Blow ptient's nose and huff, cough to clear your upper airways to mucus.This technique has three phases. Moving mucus from small airways (Unsticking), Moving mucus from small airways to medium sized airways(Collecting), Moving mucus from medium sized airways to large airways(Evacuation) Take in a deep breath.Hold the breath for three seconds.With some gentle force exhale all the air out of your lungs. Repeat three times.Do not cough untill after the third breath.
  Repeat sessions 3 times in a week for 4 almost weeks. Repeat the cycle untill you have cleared your lungs as much as possible, which should take between 20 and 45 minutes.

SUMMARY:
Chronic obstructive pulmonary disease is one of the most common life threatening disease affecting population. It is a preventable and treatable lung disease. People with COPD must work harder to breathe, which can lead to shortness of breath and/or feeling tired. Autogenic drainage (AD) works by adapting your breathing and maximizing airflow within the airways to improve ventilation and clear sputum. Segmental breathing, also referred to as localized expansion breathing, is the exercise used to improve ventilation and oxygenation. This research of randomized controlled trial will check the combined effects of segmental breathing technique and autogenic drainage technique in chronic obstructive pulmonary disease by taking sample of 40 patients through non probability convenient sampling and randomly allocating them into two groups A and B out of which A will receive both autogenic drainage and segmental breathing technique, B will receive autogenic drainage only for upto the duration of 3 days per week(20-45 min) for upto 4 weeks.Pre and post training outcomes will be measured through pulse oximeter,spirometer and BCSS.The data will be analyzed through SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 - 60 years.
* Diagnosed moderate COPD patients according to GOLD criteria.
* FEV / FVC ratio < 70 years
* Stable patients can understand written and oral english,urdu trial information.

Exclusion Criteria:

* Pregnancy, due to the Pressure on pelvic and Abdomen muscles.
* Malignant disease
* Severe (RA)
* Diagnosis of Asthma and major diseases, functionally limiting diseases, life expectancy < 3 months.
* Neurological disorders

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
SPIROMETER | baseline and fourth week
  The most used pulmonary function test is spirometry. It assesses the capacity of the lungs to breathe in and out, especially the volume and/or velocity of air that can be expelled. When evaluating breathing patterns to detect diseases including asthma, pulmonary fibrosis, cystic fibrosis, and COPD, spirometry is useful. An FEV1/FVC ratio larger than 0.70 with both FEV1 and FVC over 80% of the expected value are considered normal spirometry data. TLC exceeding 80% of the predicted value is typical in the event that lung volumes are measured. Diffusion capacity that is more than 75% of the expected value is likewise regarded as typical
PULSE OXIMETER | baseline and fourth week
  Pulse oximetry operates by shining a light through the skin at two different wavelengths_660 nm(red) and 940nm(infrared)_ and measuring the difference in light absorbance at the two wavelengths to estimate an arterial oxygen saturation
BREATHLESSNESS COUGH SPUTUM SCALE(BCSS) | baseline and fourth week
  The breathlessness cough sputum scale tool is an effective means for measuring the impact of Pulmonary rehabilitation on improving patient tolerance and self reported symptoms as the result of COPD

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Ever Care Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali RA, Obeisat SM, Tarawneh LH. Improving nursing knowledge and care for neonates with respiratory distress in Jordan. Int Nurs Rev. 2019 Sep;66(3):338-345. doi: 10.1111/inr.12510. Epub 2019 Apr 1. PMID 30937901
- [Background] Fink JB. Forced expiratory technique, directed cough, and autogenic drainage. Respir Care. 2007 Sep;52(9):1210-21; discussion 1221-3. PMID 17716387
- [Background] Zak M, Gauchez H, Boberski M, Stangret A, Kempinska-Podhorodecka A. Effectiveness of Autogenic Drainage in Improving Pulmonary Function in Patients with Cystic Fibrosis. Int J Environ Res Public Health. 2023 Feb 21;20(5):3822. doi: 10.3390/ijerph20053822. PMID 36900829